CLINICAL TRIAL: NCT00545012
Title: A 30-month Safety and Efficacy Follow-up Study With Levetiracetam at Individualized Optimal Dose in Children (4-17 Years Old at Inclusion) Suffering From Typical Absences in Childhood Absence Epilepsy (CAE) or Juvenile Absence Epilepsy (JAE)
Brief Title: A Safety and Efficacy Follow-up Study With Levetiracetam in Children (4-17 Years Old) Suffering From Absence Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N164
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Absence Seizures
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
This long-term open label follow-up trial gave pediatric subjects suffering from typical absences in CAE or JAE the opportunity to continue levetiracetam treatment after participation in the pilot study (study N162) or the double-blind study (study N163). Safety and efficacy data were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male/female 4-17 years old having participated in study N162 or in study N163
* suffering from typical absences with 3 Hz spike-wave discharges, with or without tonic-clonic seizures, in CAE or JAE
* expected reasonable benefit (efficacy and tolerability) of levetiracetam long term administration

Exclusion Criteria:

* allergy/intolerance to pyrrolidine derivatives and/or excipients
* use of > 2 concomitant antiepileptic treatment or valproate, ethosuximide or lamotrigine

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2000-05; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Continue levetiracetam treatment after participation in the pilot-study N162 or in study N163; Assess long-term safety profile and efficacy of levetiracetam

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma